CLINICAL TRIAL: NCT04526275
Title: Development of a Bruise Scale in Healthy Normal Volunteers
Brief Title: Development of Validated Bruise Scale in HNV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cearna, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CI-B002
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Bruise, Contusion
MeSH Terms: conditions — Contusions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Subjects will have a mechanically induced bruise photographed over a period of 11 days to record the healing process. Assessors will rate the bruises to develop a bruising scale.

DETAILED DESCRIPTION:
Observational study. Healthy normal volunteers will come into the clinic and have a bruise induced. The bruised area will be photographed each day through Day 11. Images will be provided to the Validator Team to rate on a 0-5 scale of severity.

The actual numbers of volunteers will be adjusted to ensure there are at least 15 images for each Grade.

The clinical site will be provided photography equipment, and study staff will be trained on photography technique to standardize the image quality and resolution across the study.

The Validator Team will review the images and categorize them in to Grades 0-5.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin type 1-3
* BMI 25 kg/m2
* Self described bruisers
* Intact skin in the target area, free of markings, blemishes and hair

Exclusion Criteria:

* Use of recreational drugs, steroids, pain medications, other homeopathic remedies, anticoagulant therapies, antiplatelet therapy
* Known history of dermal sensitivity, serious illness, hematological abnormality, impaired wound healing
* Inability to forego application of topical products in the target area
* Hair removal by laser, wax or chemicals within one week prior to Day 1
* Avoid tanning beds
* Active wound or infection in the target area
* History of keloids or hypertrophic scarring
* History of collagen or vascular disease
* History of organ transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Normal Volunteers
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-04-28 (Estimated)

PRIMARY OUTCOMES:
Bruise Healing over time | 11 days
  Record bruise images over 11 days

CONTACTS AND LOCATIONS:
Locations (1):
- Artemis Clinical Research, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be shared and published.